CLINICAL TRIAL: NCT00856856
Title: A Clinical Evaluation of the Bioabsorbable Everolimus Eluting Coronary Stent System (BVS EECSS) in the Treatment of Patients With de Novo Native Coronary Artery Lesions.
Brief Title: ABSORB Clinical Investigation, Cohort B
Acronym: ABSORB B
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-370 Cohort B
Record Dates: First submitted 2009-02-27; First posted 2009-03-06 (Estimated); Results first posted 2019-02-07 (Actual); Last update posted 2019-02-07 (Actual); Status verified 2018-01

CONDITIONS: Coronary Disease; Coronary Artery Disease; Coronary Restenosis
Keywords: Bioabsorbable; Coronary Stent; Everolimus; Drug eluting stents; Stents; Angioplasty; Coronary artery disease (CAD); Total coronary occlusion; Coronary artery restenosis; Stent thrombosis; Vascular disease; Myocardial ischemia; Coronary artery stenosis
MeSH Terms: conditions — Coronary Disease; Coronary Artery Disease; Coronary Restenosis; Vascular Diseases; Myocardial Ischemia; Coronary Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Absorb stent (Experimental): Bioabsorbable Vascular Solutions Everolimus Eluting Coronary Stent System (BVS EECSS)
  Interventions: Device: Bioabsorbable Everolimus Eluting Coronary Stent

INTERVENTIONS:
Device: Bioabsorbable Everolimus Eluting Coronary Stent — Bioabsorbable drug eluting stent implantation in the treatment of coronary artery disease

SUMMARY:
The purpose of this study is to assess the safety and performance of the BVS Everolimus Eluting Coronary Stent System (EECSS) in the treatment of patients with a maximum of two de novo native coronary artery lesions located in two different major epicardial vessels.

Currently in development at Abbott Vascular. Not available for sale in the United States.

ELIGIBILITY:
General inclusion criteria

1. Patient must be at least 18 years of age.
2. Patient is able to verbally confirm understanding of risks, benefits and treatment alternatives of receiving the BVS Everolimus Eluting CSS and he/she or his/her legally authorized representative provides written informed consent prior to any Clinical Investigation related procedure, as approved by the appropriate Ethics Committee of the respective clinical site.
3. Patient must have evidence of myocardial ischemia (e.g., stable or unstable angina, silent ischemia, positive functional study or a reversible change in the electrocardiogram (ECG) consistent with ischemia)
4. Patient must be an acceptable candidate for coronary artery bypass graft (CABG) surgery
5. Patient must agree to undergo all clinical investigation plan-required follow-up visits, angiograms, intravascular ultrasound (IVUS), Palpography (optional), optical coherence tomography (OCT) (strongly recommended), multislice computed tomography (MSCT) (optional) and coronary vasomotion (optional)
6. Patient must agree not to participate in any other clinical investigation for a period of two years following the index procedure

Angiographic Inclusion Criteria

1. Target lesion(s) must be located in a native coronary artery with visually estimated nominal vessel diameter of 3.0 mm
2. Target lesion(s) must measure ≤ 14 mm in length by visual estimation
3. Target lesion(s) must be in a major artery or branch with a visually estimated stenosis of ≥ 50% and < 100% with a TIMI flow of ≥ 1
4. If two target lesions meet the inclusion criteria they must be in different major epicardial vessels left anterior descending artery (LAD) with septal and diagonal branches, left circumflex artery (LCX) with obtuse marginal and/or ramus intermedius branches and right coronary artery (RCA) and any of its branches
5. If two target lesion(s) are being treated, each of these lesions must meet all angiographic inclusion/exclusion criteria
6. Non-Clinical Investigation, percutaneous intervention for lesions in a non-target vessel is allowed if done ≥ 90 days prior to or if planned to be done 6 months after the index procedure
7. Non-Clinical Investigation percutaneous intervention for lesion in the target vessel is allowed if done > 6 months prior to or if planned to be done 6 months after the index procedure

General Exclusion Criteria

1. Patients has had a known diagnosis of acute myocardial infarction (AMI) within 3 days preceding the index procedure and creatine kinase (CK) and CK-MB have not returned within normal limits at the time of procedure
2. The patient is currently experiencing clinical symptoms consistent with AMI
3. Patient has current unstable arrhythmias
4. Patient has a known left ventricular ejection fraction (LVEF) < 30%
5. Patient has received a heart transplant or any other organ transplant or is on a waiting list for any organ transplant
6. Patient is receiving or scheduled to receive chemotherapy for malignancy within 30 days prior to or after the procedure
7. Patient is receiving immunosuppression therapy and has known immunosuppressive or autoimmune disease (e.g. human immunodeficiency virus, systemic lupus erythematosus etc.)
8. Patient is receiving or scheduled to receive chronic anticoagulation therapy (e.g., heparin, coumadin)
9. Patient has a known hypersensitivity or contraindication to aspirin, both heparin and bivalirudin, both clopidogrel and ticlopidine, everolimus, poly (L-lactide), poly (DL-lactide) or contrast sensitivity that cannot be adequately pre-medicated
10. Elective surgery is planned within the first 6 months after the procedure that will require discontinuing either aspirin or clopidogrel
11. Patient has a platelet count < 100,000 cells/mm3 or > 700,000 cells/mm3, a white blood cell count of < 3,000 cells/mm3, or documented or suspected liver disease (including laboratory evidence of hepatitis)
12. Patient has known renal insufficiency (e.g., serum creatinine level of more than 2.5 mg/dL, or patient on dialysis)
13. Patient has a history of bleeding diathesis or coagulopathy or will refuse blood transfusions
14. Patient has had a cerebrovascular accident (CVA) or transient ischemic neurological attack (TIA) within the past six months
15. Patient has had a significant GI or urinary bleed within the past six months
16. Patient has extensive peripheral vascular disease that precludes safe 6 French sheath insertion
17. Patient has other medical illness (e.g., cancer or congestive heart failure) or known history of substance abuse (alcohol, cocaine, heroin etc.) that may cause non-compliance with the clinical investigation plan, confound the data interpretation or is associated with a limited life expectancy (i.e., less than one year)
18. Patient is already participating in another clinical investigation that has not yet reached its primary endpoint
19. Pregnant or nursing patients and those who plan pregnancy during the Clinical Investigation. (Female patients of child-bearing potential must have a negative pregnancy test done within 7 days prior to the index procedure and effective contraception must be used during participation in this Clinical Investigation)
20. Patient has received brachytherapy in any epicardial vessel (including side branches)

Angiographic Exclusion Criteria

1. Target lesion(s) meets any of the following criteria:

   1. Aorto-ostial location (within 3 mm)
   2. Left main location
   3. Located within 2 mm of the origin of the LAD or LCX
   4. Located within an arterial or saphenous vein graft or distal to a diseased (defined as vessel irregularity per angiogram and > 20% stenosed lesion, by visual estimation) arterial or saphenous vein graft
   5. Lesion involving a bifurcation ≥ 2 mm in diameter and ostial lesion > 40% stenosed by visual estimation or side branch requiring predilatation
   6. Total occlusion (TIMI flow 0), prior to wire crossing
   7. Excessive tortuosity proximal to or within the lesion
   8. Extreme angulation (≥ 90%) proximal to or within the lesion
   9. Heavy calcification
   10. Restenotic from previous intervention
2. The target vessel contains visible thrombus
3. Another clinically significant lesion is located in the same major epicardial vessel as the target lesion(s) (including side branches)
4. Patient has a high probability that a procedure other than pre-dilatation and stenting and (if necessary) post-dilatation will be required at the time of index procedure for treatment of the target vessel (e.g. atherectomy, cutting balloon or brachytherapy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2009-03; Primary Completion 2015-10 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Serruys, MD, Principal Investigator — Erasmus Heart Center, Thorax Centrum; John Ormiston, MD, Principal Investigator — Auckland City Hospital
Locations (12):
- Australia (2):
  - St. Vincent's Hospital, Melbourne, Victoria
  - Monash Heart, Melbourne
- Onze-Lieve VrouweZiekenhuis, Aalst, Belgium
- Skejby Sygehus, Aarhus, Denmark
- Institut Hospitalier Jacques Cartier, Massy, France
- Netherlands (3):
  - Catharina ZH Eindhoven, Eindhoven
  - Erasmus Medical Center, Rotterdam
  - Maasstad Ziekenhuis, Rotterdam
- New Zealand (2):
  - Auckland City Hospital, Auckland
  - Christchurch Hospital, Christchurch
- Jagiellonian University, Krakow, Poland
- Inselspital Bern, Kardiologie, Bern, Switzerland

REFERENCES:
- [Derived] Zeng Y, Cavalcante R, Collet C, Tenekecioglu E, Sotomi Y, Miyazaki Y, Katagiri Y, Asano T, Abdelghani M, Nie S, Bourantas CV, Bruining N, Onuma Y, Serruys PW. Coronary calcification as a mechanism of plaque/media shrinkage in vessels treated with bioresorbable vascular scaffold: A multimodality intracoronary imaging study. Atherosclerosis. 2018 Feb;269:6-13. doi: 10.1016/j.atherosclerosis.2017.11.002. Epub 2017 Dec 2. PMID 29247976
- [Derived] Onuma Y, Grundeken MJ, Nakatani S, Asano T, Sotomi Y, Foin N, Ng J, Okamura T, Wykrzykowska JJ, de Winter RJ, van Geuns RJ, Koolen J, Christiansen EH, Whitbourn R, McClean D, Smits P, Windecker S, Ormiston JA, Serruys PW. Serial 5-Year Evaluation of Side Branches Jailed by Bioresorbable Vascular Scaffolds Using 3-Dimensional Optical Coherence Tomography: Insights From the ABSORB Cohort B Trial (A Clinical Evaluation of the Bioabsorbable Everolimus Eluting Coronary Stent System in the Treatment of Patients With De Novo Native Coronary Artery Lesions). Circ Cardiovasc Interv. 2017 Sep;10(9):e004393. doi: 10.1161/CIRCINTERVENTIONS.116.004393. PMID 28893770
- [Derived] Zeng Y, Tateishi H, Cavalcante R, Tenekecioglu E, Suwannasom P, Sotomi Y, Collet C, Nie S, Jonker H, Dijkstra J, Radu MD, Raber L, McClean DR, van Geuns RJ, Christiansen EH, Fahrni T, Koolen J, Onuma Y, Bruining N, Serruys PW. Serial Assessment of Tissue Precursors and Progression of Coronary Calcification Analyzed by Fusion of IVUS and OCT: 5-Year Follow-Up of Scaffolded and Nonscaffolded Arteries. JACC Cardiovasc Imaging. 2017 Oct;10(10 Pt A):1151-1161. doi: 10.1016/j.jcmg.2016.11.016. Epub 2017 Mar 15. PMID 28330651
- [Derived] Onuma Y, Collet C, van Geuns RJ, de Bruyne B, Christiansen E, Koolen J, Smits P, Chevalier B, McClean D, Dudek D, Windecker S, Meredith I, Nieman K, Veldhof S, Ormiston J, Serruys PW; ABSORB Investigators. Long-term serial non-invasive multislice computed tomography angiography with functional evaluation after coronary implantation of a bioresorbable everolimus-eluting scaffold: the ABSORB cohort B MSCT substudy. Eur Heart J Cardiovasc Imaging. 2017 May 1;18(8):870-879. doi: 10.1093/ehjci/jex022. PMID 28329198
- [Derived] Serruys PW, Ormiston J, van Geuns RJ, de Bruyne B, Dudek D, Christiansen E, Chevalier B, Smits P, McClean D, Koolen J, Windecker S, Whitbourn R, Meredith I, Wasungu L, Ediebah D, Veldhof S, Onuma Y. A Polylactide Bioresorbable Scaffold Eluting Everolimus for Treatment of Coronary Stenosis: 5-Year Follow-Up. J Am Coll Cardiol. 2016 Feb 23;67(7):766-76. doi: 10.1016/j.jacc.2015.11.060. PMID 26892411
- [Derived] Ishibashi Y, Nakatani S, Sotomi Y, Suwannasom P, Grundeken MJ, Garcia-Garcia HM, Bartorelli AL, Whitbourn R, Chevalier B, Abizaid A, Ormiston JA, Rapoza RJ, Veldhof S, Onuma Y, Serruys PW. Relation Between Bioresorbable Scaffold Sizing Using QCA-Dmax and Clinical Outcomes at 1 Year in 1,232 Patients From 3 Study Cohorts (ABSORB Cohort B, ABSORB EXTEND, and ABSORB II). JACC Cardiovasc Interv. 2015 Nov;8(13):1715-26. doi: 10.1016/j.jcin.2015.07.026. PMID 26585622
- [Derived] Karanasos A, Garcia-Garcia HM, van Geuns RJ, Regar E. Fate of side-branch jailing and a malapposed platinum marker after resorption of an everolimus-eluting bioresorbable vascular scaffold: serial optical coherence tomography observations. JACC Cardiovasc Interv. 2015 Mar;8(3):e53-e54. doi: 10.1016/j.jcin.2014.10.020. No abstract available. PMID 25790767
- [Derived] Onuma Y, Serruys PW, Muramatsu T, Nakatani S, van Geuns RJ, de Bruyne B, Dudek D, Christiansen E, Smits PC, Chevalier B, McClean D, Koolen J, Windecker S, Whitbourn R, Meredith I, Garcia-Garcia HM, Veldhof S, Rapoza R, Ormiston JA. Incidence and imaging outcomes of acute scaffold disruption and late structural discontinuity after implantation of the absorb Everolimus-Eluting fully bioresorbable vascular scaffold: optical coherence tomography assessment in the ABSORB cohort B Trial (A Clinical Evaluation of the Bioabsorbable Everolimus Eluting Coronary Stent System in the Treatment of Patients With De Novo Native Coronary Artery Lesions). JACC Cardiovasc Interv. 2014 Dec;7(12):1400-11. doi: 10.1016/j.jcin.2014.06.016. PMID 25523532
- [Derived] Zhang YJ, Iqbal J, Nakatani S, Bourantas CV, Campos CM, Ishibashi Y, Cho YK, Veldhof S, Wang J, Onuma Y, Garcia-Garcia HM, Dudek D, van Geuns RJ, Serruys PW; ABSORB Cohort B Study Investigators. Scaffold and edge vascular response following implantation of everolimus-eluting bioresorbable vascular scaffold: a 3-year serial optical coherence tomography study. JACC Cardiovasc Interv. 2014 Dec;7(12):1361-9. doi: 10.1016/j.jcin.2014.06.025. Epub 2014 Nov 12. PMID 25457053
- [Derived] Muramatsu T, Onuma Y, van Geuns RJ, Chevalier B, Patel TM, Seth A, Diletti R, Garcia-Garcia HM, Dorange CC, Veldhof S, Cheong WF, Ozaki Y, Whitbourn R, Bartorelli A, Stone GW, Abizaid A, Serruys PW; ABSORB Cohort B Investigators; ABSORB EXTEND Investigators; SPIRIT FIRST Investigators; SPIRIT II Investigators; SPIRIT III Investigators; SPIRIT IV Investigators. 1-year clinical outcomes of diabetic patients treated with everolimus-eluting bioresorbable vascular scaffolds: a pooled analysis of the ABSORB and the SPIRIT trials. JACC Cardiovasc Interv. 2014 May;7(5):482-93. doi: 10.1016/j.jcin.2014.01.155. Epub 2014 Apr 16. PMID 24746650
- [Derived] Serruys PW, Onuma Y, Garcia-Garcia HM, Muramatsu T, van Geuns RJ, de Bruyne B, Dudek D, Thuesen L, Smits PC, Chevalier B, McClean D, Koolen J, Windecker S, Whitbourn R, Meredith I, Dorange C, Veldhof S, Hebert KM, Rapoza R, Ormiston JA. Dynamics of vessel wall changes following the implantation of the absorb everolimus-eluting bioresorbable vascular scaffold: a multi-imaging modality study at 6, 12, 24 and 36 months. EuroIntervention. 2014 Mar 20;9(11):1271-84. doi: 10.4244/EIJV9I11A217. PMID 24291783
- [Derived] Ormiston JA, Serruys PW, Onuma Y, van Geuns RJ, de Bruyne B, Dudek D, Thuesen L, Smits PC, Chevalier B, McClean D, Koolen J, Windecker S, Whitbourn R, Meredith I, Dorange C, Veldhof S, Hebert KM, Rapoza R, Garcia-Garcia HM. First serial assessment at 6 months and 2 years of the second generation of absorb everolimus-eluting bioresorbable vascular scaffold: a multi-imaging modality study. Circ Cardiovasc Interv. 2012 Oct;5(5):620-32. doi: 10.1161/CIRCINTERVENTIONS.112.971549. Epub 2012 Oct 9. PMID 23048057
- [Derived] Gutierrez-Chico JL, Gijsen F, Regar E, Wentzel J, de Bruyne B, Thuesen L, Ormiston J, McClean DR, Windecker S, Chevalier B, Dudek D, Whitbourn R, Brugaletta S, Onuma Y, Serruys PW. Differences in neointimal thickness between the adluminal and the abluminal sides of malapposed and side-branch struts in a polylactide bioresorbable scaffold: evidence in vivo about the abluminal healing process. JACC Cardiovasc Interv. 2012 Apr;5(4):428-35. doi: 10.1016/j.jcin.2011.12.015. PMID 22516401
- [Derived] Brugaletta S, Radu MD, Garcia-Garcia HM, Heo JH, Farooq V, Girasis C, van Geuns RJ, Thuesen L, McClean D, Chevalier B, Windecker S, Koolen J, Rapoza R, Miquel-Hebert K, Ormiston J, Serruys PW. Circumferential evaluation of the neointima by optical coherence tomography after ABSORB bioresorbable vascular scaffold implantation: can the scaffold cap the plaque? Atherosclerosis. 2012 Mar;221(1):106-12. doi: 10.1016/j.atherosclerosis.2011.12.008. Epub 2011 Dec 13. PMID 22209268
- [Derived] Gutierrez-Chico JL, Radu MD, Diletti R, Sheehy A, Kossuth MB, Oberhauser JP, Glauser T, Harrington J, Rapoza RJ, Onuma Y, Serruys PW. Spatial distribution and temporal evolution of scattering centers by optical coherence tomography in the poly(L-lactide) backbone of a bioresorbable vascular scaffold. Circ J. 2012;76(2):342-50. doi: 10.1253/circj.cj-11-0726. Epub 2011 Nov 19. PMID 22104034
- [Derived] Serruys PW, Onuma Y, Dudek D, Smits PC, Koolen J, Chevalier B, de Bruyne B, Thuesen L, McClean D, van Geuns RJ, Windecker S, Whitbourn R, Meredith I, Dorange C, Veldhof S, Hebert KM, Sudhir K, Garcia-Garcia HM, Ormiston JA. Evaluation of the second generation of a bioresorbable everolimus-eluting vascular scaffold for the treatment of de novo coronary artery stenosis: 12-month clinical and imaging outcomes. J Am Coll Cardiol. 2011 Oct 4;58(15):1578-88. doi: 10.1016/j.jacc.2011.05.050. PMID 21958884
- [Derived] Gomez-Lara J, Radu M, Brugaletta S, Farooq V, Diletti R, Onuma Y, Windecker S, Thuesen L, McClean D, Koolen J, Whitbourn R, Dudek D, Smits PC, Regar E, Veldhof S, Rapoza R, Ormiston JA, Garcia-Garcia HM, Serruys PW. Serial analysis of the malapposed and uncovered struts of the new generation of everolimus-eluting bioresorbable scaffold with optical coherence tomography. JACC Cardiovasc Interv. 2011 Sep;4(9):992-1001. doi: 10.1016/j.jcin.2011.03.020. PMID 21939939
- [Derived] Gomez-Lara J, Brugaletta S, Farooq V, van Geuns RJ, De Bruyne B, Windecker S, McClean D, Thuesen L, Dudek D, Koolen J, Whitbourn R, Smits PC, Chevalier B, Morel MA, Dorange C, Veldhof S, Rapoza R, Garcia-Garcia HM, Ormiston JA, Serruys PW. Angiographic geometric changes of the lumen arterial wall after bioresorbable vascular scaffolds and metallic platform stents at 1-year follow-up. JACC Cardiovasc Interv. 2011 Jul;4(7):789-99. doi: 10.1016/j.jcin.2011.04.009. PMID 21777888
- [Derived] Gutierrez-Chico JL, Serruys PW, Girasis C, Garg S, Onuma Y, Brugaletta S, Garcia-Garcia H, van Es GA, Regar E. Quantitative multi-modality imaging analysis of a fully bioresorbable stent: a head-to-head comparison between QCA, IVUS and OCT. Int J Cardiovasc Imaging. 2012 Mar;28(3):467-78. doi: 10.1007/s10554-011-9829-y. Epub 2011 Feb 26. PMID 21359517
- [Derived] Serruys PW, Onuma Y, Ormiston JA, de Bruyne B, Regar E, Dudek D, Thuesen L, Smits PC, Chevalier B, McClean D, Koolen J, Windecker S, Whitbourn R, Meredith I, Dorange C, Veldhof S, Miquel-Hebert K, Rapoza R, Garcia-Garcia HM. Evaluation of the second generation of a bioresorbable everolimus drug-eluting vascular scaffold for treatment of de novo coronary artery stenosis: six-month clinical and imaging outcomes. Circulation. 2010 Nov 30;122(22):2301-12. doi: 10.1161/CIRCULATIONAHA.110.970772. Epub 2010 Nov 15. PMID 21098436
- [Derived] Gomez-Lara J, Garcia-Garcia HM, Onuma Y, Garg S, Regar E, De Bruyne B, Windecker S, McClean D, Thuesen L, Dudek D, Koolen J, Whitbourn R, Smits PC, Chevalier B, Dorange C, Veldhof S, Morel MA, de Vries T, Ormiston JA, Serruys PW. A comparison of the conformability of everolimus-eluting bioresorbable vascular scaffolds to metal platform coronary stents. JACC Cardiovasc Interv. 2010 Nov;3(11):1190-8. doi: 10.1016/j.jcin.2010.07.016. PMID 21087756
- [Derived] Okamura T, Onuma Y, Garcia-Garcia HM, Regar E, Wykrzykowska JJ, Koolen J, Thuesen L, Windecker S, Whitbourn R, McClean DR, Ormiston JA, Serruys PW; ABSORB Cohort B Investigators. 3-Dimensional optical coherence tomography assessment of jailed side branches by bioresorbable vascular scaffolds: a proposal for classification. JACC Cardiovasc Interv. 2010 Aug;3(8):836-44. doi: 10.1016/j.jcin.2010.05.011. PMID 20723856
- See also: Absorb, cohort A — http://www.clinicaltrials.gov/ct2/show/NCT00300131?term=absorb&rank=1

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total of 101 patients (intent to treat patient population [ITT]) were enrolled in the ABSORB Cohort B study at 12 clinical sites in Europe/Australia/New Zealand between March 19, 2009 and November 6, 2009. Only for assessing imaging outcomes at different follow-up periods, subjects were divided into Group 1 (n = 45) & Group 2 (n = 56).
Pre-assignment Details: ITT population were assessed for all clinical endpoints. For imaging outcomes,Group 1 (n=45) patients were followed up at 180 days, 2 & 5 years; while Group 2 (n=56) patients at 1, 3 & 5 years. Therefore, data related to imaging outcomes are available only for Group 1 at 180 days, 2 & 5 years timeframe & only for Group 2 at 1, 3 & 5 years timeframe
Groups:
- Absorb BVS: Bioabsorbable Vascular Solutions Everolimus Eluting Coronary Stent System (BVS EECSS)
  Bioabsorbable Everolimus Eluting Coronary Stent: Bioabsorbable drug eluting stent implantation in the treatment of coronary artery disease.
  Investigational devices available for the study were the Absorb BVS with a diameter of 3.0 mm and length of 18 mm. A total of 249 Absorb BVS were received at 12 investigational sites in the ABSORB Cohort B clinical study. Of the 249 devices received by the study sites, 102 were implanted in patients and 147 were returned to the sponsor.
Period: Baseline
Arm/Group | Absorb BVS
Started | 101
Completed | 101
Not Completed | 0
Period: 30-day Clinical Follow-up
Arm/Group | Absorb BVS
Started | 101
Completed | 101
Not Completed | 0
Period: 180-day Clinical Follow-up
Arm/Group | Absorb BVS
Started | 101
Completed | 101
Not Completed | 0
Period: 270-day Clinical Follow-up
Arm/Group | Absorb BVS
Started | 101
Completed | 101
Not Completed | 0
Period: 1-year Clinical Follow-up
Arm/Group | Absorb BVS
Started | 101
Completed | 101
Not Completed | 0
Period: 2-year Clinical Follow-up
Arm/Group | Absorb BVS
Started | 101
Completed | 100
Not Completed | 1
Not completed — Lost to Follow-up | 1
Period: 3-year Clinical Follow-up
Arm/Group | Absorb BVS
Started | 100
Completed | 100
Not Completed | 0
Period: 4-year Clinical Follow-up
Arm/Group | Absorb BVS
Started | 100
Completed | 99
Not Completed | 1
Not completed — Missed visit | 1
Period: 5-year Clinical Follow-up
Arm/Group | Absorb BVS
Started | 100
Completed | 100 (One patient missed the 4-year clinical follow-up but returned at 5 year.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The patient demographics for the full Cohort B 101 patients (Group 1, 45 patients and Group 2, 56 patients) are described.
Groups:
- Absorb BVS: Bioabsorbable Vascular Solutions Everolimus Eluting Coronary Stent System (BVS EECSS)
  Bioabsorbable Everolimus Eluting Coronary Stent: Bioabsorbable drug eluting stent implantation in the treatment of coronary artery disease.
  Investigational devices available for the study were the Absorb BVS with a diameter of 3.0 mm and length of 18 mm. A total of 249 Absorb BVS were received at twelve investigational sites in the ABSORB Cohort B clinical study. Of the 249 devices received by the study sites, 102 were implanted in patients and 147 were returned to the sponsor.
Arm/Group | Absorb BVS
Number analyzed (Participants) | 101
Age, Continuous [Mean (Full Range); unit: years] | 62.3 [60.4 to 64.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 73
Region of Enrollment [Number; unit: participants]
  New Zealand | 14
  Netherlands | 30
  Belgium | 14
  Poland | 13
  Denmark | 12
  France | 8
  Australia | 4
  Switzerland | 6

OUTCOME MEASURES:

1. Primary Outcome: Hierarchical Major Adverse Cardiac Event (MACE)
Description: Major adverse cardiac events (MACE) is defined as the composite of cardiac death, all myocardial infarction,and clinically indicated target lesion revascularization (CI-TLR).
Time Frame: 30 days
Population: Analysis population includes both Group 1 (n=45) and Group 2 (n=56) patients. Intent-to-treat (ITT) population.
Measure: Number; unit: percentage of participants
Arm/Group | Absorb BVS
Number analyzed (Participants) | 101
percentage of participants | 2.0

2. Primary Outcome: Hierarchical Major Adverse Cardiac Event (MACE)
Description: as for outcome 1
Time Frame: 1 year
Population: Analysis population includes both Group 1 (n=45) and Group 2 (n=56) patients. Intent-to-treat (ITT) population.
Measure: Number; unit: percentage of participants
Arm/Group | Absorb BVS
Number analyzed (Participants) | 101
percentage of participants | 6.9

3. Primary Outcome: In-scaffold Late Loss: In-scaffold MLD Post-procedure - In-scaffold MLD at 180 Days
Description: In-scaffold Late Loss: in-scaffold MLD post-procedure - in-scaffold MLD at follow-up.
Time Frame: 180 days
Population: In Cohort B, Group 1. Intent-to-treat (ITT) population. The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: Millimeter
Units Other Than Participants: Target lesions
Groups:
- Absorb BVS: Bioabsorbable Vascular Solutions Everolimus Eluting Coronary Stent System (BVS EECSS).
  Bioabsorbable Everolimus Eluting Coronary Stent: Bioabsorbable drug eluting stent implantation in the treatment of coronary artery disease.
  Investigational devices available for the study were the Absorb BVS with a diameter of 3.0 mm and length of 18 mm.
  Cohort B patients were split into Group 1 having imaging follow-up at 180 days and 2 years and Group 2 having imaging follow-up at 1 year and 3 years.
Arm/Group | Absorb BVS
Number analyzed (Participants) | 42
Number analyzed (Target lesions) | 42
Millimeter | 0.19 (0.18)

4. Primary Outcome: In-scaffold Late Loss: In-scaffold MLD Post-procedure - In-scaffold MLD at 1 Year
Description: In-scaffold Late Loss: in-scaffold MLD post-procedure - in-scaffold MLD at follow-up
Time Frame: 1 year
Population: In Cohort B, Group 2. Intent-to-treat (ITT) population. The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: Millimeter
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 56
Number analyzed (Target lesions) | 57
Millimeter | 0.27 (0.32)

5. Secondary Outcome: Clinical Device Success (Per Lesion)
Description: Successful delivery and deployment of the Clinical Investigation scaffold at the intended target lesion and successful withdrawal of the scaffold delivery system with attainment of final residual stenosis of less than 50% of the target lesion by QCA (by visual estimation if QCA unavailable). Standard pre-dilation catheters and post-dilatation catheters (if applicable) may be used. Bailout patients will be included as device success only if the above criteria for clinical device are met.
Time Frame: On day 0 (the day of procedure)
Population: Analysis population includes both Group 1 (n=45) and Group 2 (n=56) patients. Intent-to-treat (ITT) population.
Measure: Number; unit: percentage of lesions
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 101
Number analyzed (Target lesions) | 102
percentage of lesions | 100.0

6. Secondary Outcome: Clinical Procedure Success (Per Patient)
Description: Successful delivery and deployment of the Clinical Investigation scaffold at the intended target lesion and successful withdrawal of the scaffold delivery system with attainment of final residual stenosis of less than 50% of the target lesion by QCA (by visual estimation if QCA unavailable) and/or using any adjunctive device without the occurrence of ischemia-driven major adverse cardiac event (MACE) during the hospital stay with a maximum of first seven days post index procedure.
Time Frame: On day 0 (the day of procedure)
Population: Analysis population includes both Group 1 (n=45) and Group 2 (n=56) patients. Intent-to-treat (ITT) population.
Measure: Number; unit: percentage of participants
Groups:
- ABSORB Stent: Bioabsorbable Vascular Solutions Everolimus Eluting Coronary Stent System (BVS EECSS)
  Bioabsorbable Everolimus Eluting Coronary Stent: Bioabsorbable drug eluting stent implantation in the treatment of coronary artery disease.
  Investigational devices available for the study were the Absorb BVS with a diameter of 3.0 mm and length of 18 mm. A total of 249 Absorb BVS were received at twelve investigational sites in the ABSORB Cohort B clinical study. Of the 249 devices received by the study sites, 102 were implanted in patients and 147 were returned to the sponsor.
Arm/Group | ABSORB Stent
Number analyzed (Participants) | 101
percentage of participants | 98.0

7. Secondary Outcome: Hierarchical Major Adverse Cardiac Event (MACE)
Description: as for outcome 1
Time Frame: 180 days
Population: Analysis population includes both Group 1 (n=45) and Group 2 (n=56) patients. Intent-to-treat (ITT) population.
Measure: Number; unit: percentage of participants
Arm/Group | Absorb BVS
Number analyzed (Participants) | 101
percentage of participants | 5.0

8. Secondary Outcome: Hierarchical Major Adverse Cardiac Event (MACE)
Description: as for outcome 1
Time Frame: 270 days
Population: Analysis population includes both Group 1 (n=45) and Group 2 (n=56) patients. Intent-to-treat (ITT) population.
Measure: Number; unit: percentage of participants
Arm/Group | Absorb BVS
Number analyzed (Participants) | 101
percentage of participants | 5.0

9. Secondary Outcome: Hierarchical Major Adverse Cardiac Event (MACE)
Description: as for outcome 1
Time Frame: 2 years
Population: Intent-to-treat (ITT) population. Analysis population includes both Group 1 (n=44) and Group 2 (n=56) patients. One patient (Group 1) lost to follow-up at 2-year follow-up period.
Measure: Number; unit: percentage of participants
Arm/Group | Absorb BVS
Number analyzed (Participants) | 100
percentage of participants | 9.0

10. Secondary Outcome: Hierarchical Major Adverse Cardiac Event (MACE)
Description: as for outcome 1
Time Frame: 3 years
Population: Intent-to-treat (ITT) population. Analysis population includes both Group 1 (n=44) and Group 2 (n=56) patients. One patient (Group 1) lost to follow-up at 3-year follow-up period.
Measure: Number; unit: percentage of participants
Arm/Group | Absorb BVS
Number analyzed (Participants) | 100
percentage of participants | 10.0

11. Secondary Outcome: Hierarchical Major Adverse Cardiac Event (MACE)
Description: as for outcome 1
Time Frame: 4 years
Population: Analysis population includes both Group 1 (n=43) and Group 2 (n=56) patients. Two patients (Group 1) lost to follow-up at 4-year follow-up period. Intent-to-treat (ITT) population.
Measure: Number; unit: percentage of participants
Arm/Group | Absorb BVS
Number analyzed (Participants) | 99
percentage of participants | 10.1

12. Secondary Outcome: Hierarchical Major Adverse Cardiac Event (MACE)
Description: as for outcome 1
Time Frame: 5 years
Population: Analysis population includes both Group 1 (n=44) and Group 2 (n=56) patients. One patient from Group 1 population had lost-to-follow-up. Where as,1 patient (Group 1) missed the 4-year follow up but returned for the 5-year follow up. Intent-to-treat (ITT) population.
Measure: Number; unit: percentage of participants
Arm/Group | Absorb BVS
Number analyzed (Participants) | 100
percentage of participants | 11.0

13. Secondary Outcome: Hierarchical Target Vessel Failure (TVF)
Description: Target Vessel Failure (TVF) is the composite of Cardiac Death, Myocardial infarction (MI) or Ischemic-Driven Target Vessel Revascularization (ID-TVR).
Time Frame: 30 days
Population: Intent-to-treat (ITT) population. Analysis population includes both Group 1 (n=45) and Group 2 (n=56) patients.
Measure: Number; unit: percentage of participants
Arm/Group | Absorb BVS
Number analyzed (Participants) | 101
percentage of participants | 2.0

14. Secondary Outcome: Hierarchical Target Vessel Failure (TVF)
Description: as for outcome 13
Time Frame: 180 days
Population: Intent-to-treat (ITT) population. Analysis population includes both Group 1 (n=45) and Group 2 (n=56) patients.
Measure: Number; unit: Percentage of participants
Arm/Group | ABSORB Stent
Number analyzed (Participants) | 101
Percentage of participants | 5.0

15. Secondary Outcome: Hierarchical Target Vessel Failure (TVF)
Description: as for outcome 13
Time Frame: 270 days
Population: Intent-to-treat (ITT) population. Analysis population includes both Group 1 (n=45) and Group 2 (n=56) patients.
Measure: Number; unit: Percentage of participants
Arm/Group | Absorb Stent
Number analyzed (Participants) | 101
Percentage of participants | 5.0

16. Secondary Outcome: Hierarchical Target Vessel Failure (TVF)
Description: as for outcome 13
Time Frame: 1 year
Population: Intent-to-treat (ITT) population. Analysis population includes both Group 1 (n=45) and Group 2 (n=56) patients.
Measure: Number; unit: percentage of participants
Arm/Group | Absorb BVS
Number analyzed (Participants) | 101
percentage of participants | 6.9

17. Secondary Outcome: Hierarchical Target Vessel Failure (TVF)
Description: as for outcome 13
Time Frame: 2 years
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | Absorb BVS
Number analyzed (Participants) | 100
percentage of participants | 11.0

18. Secondary Outcome: Hierarchical Target Vessel Failure (TVF)
Description: as for outcome 13
Time Frame: 3 years
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Absorb BVS
Number analyzed (Participants) | 100
percentage of participants | 13.0

19. Secondary Outcome: Hierarchical Target Vessel Failure (TVF)
Description: as for outcome 13
Time Frame: 4 years
Population: Intent-to-treat (ITT) population. Analysis population includes both Group 1 (n=43) and Group 2 (n=56) patients. Two patients (Group 1) lost to follow-up at 4-year follow-up period.
Measure: Number; unit: percentage of participants
Arm/Group | Absorb BVS
Number analyzed (Participants) | 99
percentage of participants | 13.1

20. Secondary Outcome: Hierarchical Target Vessel Failure (TVF)
Description: as for outcome 13
Time Frame: 5 years
Population: Intent-to-treat (ITT) population. Analysis population includes both Group 1 (n=44) and Group 2 (n=56) patients. One patient from Group 1 population had lost-to-follow-up. Where as,1 patient (Group 1) missed the 4-year follow up but returned for the 5-year follow up.
Measure: Number; unit: percentage of participants
Arm/Group | Absorb BVS
Number analyzed (Participants) | 100
percentage of participants | 14.0

21. Secondary Outcome: Ischemia Driven Target Lesion Revascularization (ID-TLR)
Description: ID-TLR is defined as the revascularization at the target lesion associated with any of the following:
  * Positive functional ischemia study
  * Ischemic symptoms and angiographic minimal lumen diameter stenosis ≥ 50% by core laboratory quantitative coronary angiography (QCA)
  * Revascularization of a target lesion with diameter stenosis ≥ 70% by core laboratory QCA without either ischemic symptoms or a positive functional study.
Time Frame: 30 days
Population: Intent-to-treat (ITT) population. Analysis population includes both Group 1 (n=45) and Group 2 (n=56) patients.
Measure: Number; unit: percentage of participants
Arm/Group | Absorb BVS
Number analyzed (Participants) | 101
percentage of participants | 0

22. Secondary Outcome: Ischemia Driven Target Lesion Revascularization (ID-TLR)
Description: as for outcome 21
Time Frame: 180 days
Population: Intent-to-treat (ITT) population. Analysis population includes both Group 1 (n=45) and Group 2 (n=56) patients.
Measure: Number; unit: Percentage of participants
Arm/Group | Absorb BVS
Number analyzed (Participants) | 101
Percentage of participants | 2.0

23. Secondary Outcome: Ischemia Driven Target Lesion Revascularization (ID-TLR)
Description: as for outcome 21
Time Frame: 270 days
Population: Intent-to-treat (ITT) population. Analysis population includes both Group 1 (n=45) and Group 2 (n=56) patients.
Measure: Number; unit: Percentage of participants
Arm/Group | Absorb BVS
Number analyzed (Participants) | 101
Percentage of participants | 2.0

24. Secondary Outcome: Ischemia Driven Target Lesion Revascularization (ID-TLR)
Description: as for outcome 21
Time Frame: 1 year
Population: Intent-to-treat (ITT) population. Analysis population includes both Group 1 (n=45) and Group 2 (n=56) patients.
Measure: Number; unit: percentage of participants
Arm/Group | Absorb BVS
Number analyzed (Participants) | 101
percentage of participants | 4.0

25. Secondary Outcome: Ischemia Driven Target Lesion Revascularization (ID-TLR)
Description: as for outcome 21
Time Frame: 2 years
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | Absorb BVS
Number analyzed (Participants) | 100
percentage of participants | 6.0

26. Secondary Outcome: Ischemia Driven Target Lesion Revascularization (ID-TLR)
Description: as for outcome 21
Time Frame: 3 years
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Absorb BVS
Number analyzed (Participants) | 100
percentage of participants | 7.0

27. Secondary Outcome: Ischemia Driven Target Lesion Revascularization (ID-TLR)
Description: as for outcome 21
Time Frame: 4 years
Population: as for outcome 19
Measure: Number; unit: percentage of participants
Arm/Group | Absorb BVS
Number analyzed (Participants) | 99
percentage of participants | 7.1

28. Secondary Outcome: Ischemia Driven Target Lesion Revascularization (ID-TLR)
Description: as for outcome 21
Time Frame: 5 years
Population: as for outcome 20
Measure: Number; unit: percentage of participants
Arm/Group | Absorb BVS
Number analyzed (Participants) | 100
percentage of participants | 8.0

29. Secondary Outcome: Ischemia Driven Target Vessel Revascularization (ID-TVR)
Description: ID-TVR is the revascularization in the target vessel associated with any of the following:
  * Positive functional ischemia study
  * Ischemic symptoms and an angiographic minimal lumen diameter stenosis ≥ 50% by core laboratory quantitative coronary angiography (QCA)
  * Revascularization of a target vessel with diameter stenosis ≥ 70% by core laboratory QCA without either ischemic symptoms or a positive functional study.
Time Frame: 30 days
Population: Intent-to-treat (ITT) population. Analysis population includes both Group 1 (n=45) and Group 2 (n=56) patients.
Measure: Number; unit: Percentage of participants
Arm/Group | Absorb BVS
Number analyzed (Participants) | 101
Percentage of participants | 0.0

30. Secondary Outcome: Ischemia Driven Target Vessel Revascularization (ID-TVR)
Description: as for outcome 29
Time Frame: 180 days
Population: Intent-to-treat (ITT) population. Analysis population includes both Group 1 (n=45) and Group 2 (n=56) patients.
Measure: Number; unit: Percentage of participants
Arm/Group | Absorb BVS
Number analyzed (Participants) | 101
Percentage of participants | 2.0

31. Secondary Outcome: Ischemia Driven Target Vessel Revascularization (ID-TVR)
Description: as for outcome 29
Time Frame: 270 days
Population: Intent-to-treat (ITT) population. Analysis population includes both Group 1 (n=45) and Group 2 (n=56) patients.
Measure: Number; unit: Percentage of participants
Arm/Group | Absorb BVS
Number analyzed (Participants) | 101
Percentage of participants | 2.0

32. Secondary Outcome: Ischemia Driven Target Vessel Revascularization (ID-TVR)
Description: as for outcome 29
Time Frame: 1 year
Population: Intent-to-treat (ITT) population. Analysis population includes both Group 1 (n=45) and Group 2 (n=56) patients.
Measure: Number; unit: Percentage of participants
Arm/Group | Absorb BVS
Number analyzed (Participants) | 101
Percentage of participants | 4.0

33. Secondary Outcome: Ischemia Driven Target Vessel Revascularization (ID-TVR)
Description: as for outcome 29
Time Frame: 2 years
Population: as for outcome 9
Measure: Number; unit: Percentage of participants
Arm/Group | Absorb BVS
Number analyzed (Participants) | 100
Percentage of participants | 8.0

34. Secondary Outcome: Ischemia Driven Target Vessel Revascularization (ID-TVR)
Description: as for outcome 29
Time Frame: 3 years
Population: as for outcome 10
Measure: Number; unit: Percentage of participants
Arm/Group | Absorb BVS
Number analyzed (Participants) | 100
Percentage of participants | 10.0

35. Secondary Outcome: Ischemia Driven Target Vessel Revascularization (ID-TVR)
Description: as for outcome 29
Time Frame: 4 years
Population: Intent-to-treat (ITT) population. Analysis population includes both Group 1 (n=43) and Group 2 (n=56) patients. Two patient (Group 1) lost to follow-up at 4-year follow-up period.
Measure: Number; unit: Percentage of participants
Arm/Group | Absorb BVS
Number analyzed (Participants) | 99
Percentage of participants | 10.0

36. Secondary Outcome: Ischemia Driven Target Vessel Revascularization (ID-TVR)
Description: as for outcome 29
Time Frame: 5 years
Population: as for outcome 20
Measure: Number; unit: Percentage of participants
Arm/Group | Absorb BVS
Number analyzed (Participants) | 100
Percentage of participants | 11.0

37. Secondary Outcome: Cardiac Death
Description: Cardiac death is defined as any death in which a cardiac cause cannot be excluded.
  (This includes but is not limited to acute myocardial infarction, cardiac perforation/pericardial tamponade, arrhythmia or conduction abnormality, cerebrovascular accident within 30 days of the procedure or cerebrovascular accident suspected of being related to the procedure, death due to complication of the procedure, including bleeding, vascular repair, transfusion reaction, or bypass surgery.)
Time Frame: 30 days
Population: Intent-to-treat (ITT) population. Analysis population includes both Group 1 (n=45) and Group 2 (n=56) patients.
Measure: Number; unit: percentage of participants
Arm/Group | ABSORB Stent
Number analyzed (Participants) | 101
percentage of participants | 0

38. Secondary Outcome: Cardiac Death
Description: as for outcome 37
Time Frame: 1 year
Population: Intent-to-treat (ITT) population. Analysis population includes both Group 1 (n=45) and Group 2 (n=56) patients.
Measure: Number; unit: percentage of participants
Arm/Group | ABSORB Stent
Number analyzed (Participants) | 101
percentage of participants | 0

39. Secondary Outcome: Cardiac Death
Description: as for outcome 37
Time Frame: 2 years
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | ABSORB Stent
Number analyzed (Participants) | 100
percentage of participants | 0

40. Secondary Outcome: Cardiac Death
Description: as for outcome 37
Time Frame: 3 years
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | ABSORB Stent
Number analyzed (Participants) | 100
percentage of participants | 0

41. Secondary Outcome: Cardiac Death
Description: as for outcome 37
Time Frame: 4 years
Population: as for outcome 19
Measure: Number; unit: percentage of participants
Arm/Group | ABSORB Stent
Number analyzed (Participants) | 99
percentage of participants | 0

42. Secondary Outcome: Cardiac Death
Description: as for outcome 37
Time Frame: 5 years
Population: as for outcome 20
Measure: Number; unit: percentage of participants
Arm/Group | ABSORB Stent
Number analyzed (Participants) | 100
percentage of participants | 0

43. Secondary Outcome: Myocardial Infarction
Description: Myocardial Infarction (MI):
  * Q wave MI: Development of new, pathological Q wave on the ECG.
  * Non-Q wave MI: Elevation of Creatine kinase (CK) levels to ≥ two times the upper limit of normal (ULN) with elevated CK-MB in the absence of new pathological Q waves.
Time Frame: 30 days
Population: Intent-to-treat (ITT) population. Analysis population includes both Group 1 (n=45) and Group 2 (n=56) patients.
Measure: Number; unit: percentage of participants
Arm/Group | ABSORB Stent
Number analyzed (Participants) | 101
percentage of participants | 2.0

44. Secondary Outcome: Myocardial Infarction
Description: Myocardial Infarction (MI):
  * Q wave MI: Development of new, pathological Q wave on the ECG.
  * Non-Q wave MI: Elevation of CK levels to ≥ two times the upper limit of normal (ULN) with elevated CK-MB in the absence of new pathological Q waves.
Time Frame: 1 year
Population: Intent-to-treat (ITT) population. Analysis population includes both Group 1 (n=45) and Group 2 (n=56) patients.
Measure: Number; unit: percentage of participants
Arm/Group | ABSORB Stent
Number analyzed (Participants) | 101
percentage of participants | 3.0

45. Secondary Outcome: Myocardial Infarction
Description: as for outcome 44
Time Frame: 2 years
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | ABSORB Stent
Number analyzed (Participants) | 100
percentage of participants | 3.0

46. Secondary Outcome: Myocardial Infarction
Description: as for outcome 44
Time Frame: 3 years
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | ABSORB Stent
Number analyzed (Participants) | 100
percentage of participants | 3.0

47. Secondary Outcome: Myocardial Infarction
Description: as for outcome 44
Time Frame: 4 years
Population: as for outcome 19
Measure: Number; unit: percentage of participants
Arm/Group | ABSORB Stent
Number analyzed (Participants) | 99
percentage of participants | 3.0

48. Secondary Outcome: Myocardial Infarction
Description: as for outcome 44
Time Frame: 5 years
Population: as for outcome 20
Measure: Number; unit: percentage of participants
Arm/Group | ABSORB Stent
Number analyzed (Participants) | 100
percentage of participants | 3.0

49. Secondary Outcome: Scaffold Thrombosis
Description: Scaffold thrombosis will be categorized as acute (≤ 1day), subacute (>1day ≤ 30 days) and late (>30 days) and will be defined as any of the following:
  * Clinical presentation of acute coronary syndrome with angiographic evidence of scaffold thrombosis (angiographic appearance of thrombus within or adjacent to a previously treated target lesion)
  * In the absence of angiography, any unexplained death, or acute MI (ST segment elevation or new Q-wave)* in the distribution of the target lesion within 30 days *(Non-specific ST /T changes and cardiac enzyme elevations do not suffice)
  Any thromboses that occur less than 30 days after the index procedure will not be counted as restenosis.
Time Frame: 30 days
Population: Intent-to-treat (ITT) population. Analysis population includes both Group 1 (n=45) and Group 2 (n=56) patients.
Measure: Number; unit: percentage of participants
Arm/Group | ABSORB Stent
Number analyzed (Participants) | 101
percentage of participants | 0

50. Secondary Outcome: Scaffold Thrombosis
Description: as for outcome 49
Time Frame: 1 year
Population: Intent-to-treat (ITT) population. Analysis population includes both Group 1 (n=45) and Group 2 (n=56) patients.
Measure: Number; unit: percentage of participants
Arm/Group | Absorb BVS
Number analyzed (Participants) | 101
percentage of participants | 0

51. Secondary Outcome: Scaffold Thrombosis
Description: as for outcome 49
Time Frame: 2 years
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | Absorb BVS
Number analyzed (Participants) | 100
percentage of participants | 0

52. Secondary Outcome: Scaffold Thrombosis
Description: as for outcome 49
Time Frame: 3 years
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Absorb BVS
Number analyzed (Participants) | 100
percentage of participants | 0

53. Secondary Outcome: Scaffold Thrombosis
Description: as for outcome 49
Time Frame: 4 years
Population: as for outcome 19
Measure: Number; unit: percentage of participants
Arm/Group | Absorb BVS
Number analyzed (Participants) | 99
percentage of participants | 0

54. Secondary Outcome: Scaffold Thrombosis
Description: as for outcome 49
Time Frame: 5 years
Population: as for outcome 20
Measure: Number; unit: percentage of participants
Arm/Group | Absorb BVS
Number analyzed (Participants) | 100
percentage of participants | 0

55. Secondary Outcome: In-scaffold Late Loss (LL): In-scaffold MLD Post-procedure - In-scaffold MLD at 2 Years
Description: In-scaffold Late Loss: in-scaffold MLD post-procedure - in-scaffold MLD at follow-up.
Time Frame: 2 years
Population: ITT population. In Cohort B, Group 1. The number of participants analyzed include subjects who had available follow-up data at that time frame.
Measure: Mean (Standard Deviation); unit: Millimeter
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 38
Number analyzed (Target lesions) | 38
Millimeter | 0.27 (0.19)

56. Secondary Outcome: In-scaffold Late Loss (LL): In-scaffold MLD Post-procedure - In-scaffold MLD at 3 Years
Description: In-scaffold Late Loss: in-scaffold MLD post-procedure - in-scaffold MLD at follow-up.
Time Frame: 3 years
Population: Intent-to-treat (ITT) population. In Cohort B, Group 2. The number of participants analyzed include subjects who had available follow-up data at that time frame.
Measure: Mean (Standard Deviation); unit: Millimeter
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 50
Number analyzed (Target lesions) | 51
Millimeter | 0.29 (0.43)

57. Secondary Outcome: In-scaffold Late Loss (LL): In-scaffold MLD Post-procedure - In-scaffold MLD at 5 Years
Description: In-scaffold Late Loss: in-scaffold MLD post-procedure - in-scaffold MLD at follow-up.
Time Frame: 5 years
Population: Intent-to-treat (ITT) population. Cohort B, Group 1 and Group 2. The number of participants analyzed include subjects who had available follow-up data at that time frame.
Measure: Mean (Standard Deviation); unit: Millimeter
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 62
Number analyzed (Target lesions) | 63
Millimeter | 0.26 (0.42)

58. Secondary Outcome: Proximal Late Loss: Proximal MLD Post-procedure - Proximal MLD at 180 Days
Description: Proximal Late Loss: proximal MLD post-procedure - proximal MLD at follow-up (proximal defined as within 5 mm of healthy tissue proximal to scaffold placement).
Time Frame: 180 days
Population: Intent-to-treat (ITT) population. In Cohort B, Group 1. The number of participants analyzed include subjects who had available follow-up data at that time frame.
Measure: Mean (Standard Deviation); unit: Millimeter
Units Other Than Participants: Target lesions
Groups:
- Absorb BVS: Bioabsorbable Vascular Solutions Everolimus Eluting Coronary Stent System (BVS EECSS)
  Bioabsorbable Everolimus Eluting Coronary Stent: Bioabsorbable drug eluting stent implantation in the treatment of coronary artery disease
Arm/Group | Absorb BVS
Number analyzed (Participants) | 42
Number analyzed (Target lesions) | 42
Millimeter | 0.07 (0.27)

59. Secondary Outcome: Proximal Late Loss: Proximal MLD Post-procedure - Proximal MLD at 1 Year
Description: as for outcome 58
Time Frame: 1 year
Population: as for outcome 56
Measure: Mean (Standard Deviation); unit: Millimeter
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 47
Number analyzed (Target lesions) | 48
Millimeter | 0.12 (0.29)

60. Secondary Outcome: Proximal Late Loss: Proximal MLD Post-procedure - Proximal MLD at 2 Years
Description: as for outcome 58
Time Frame: 2 years
Population: as for outcome 58
Measure: Mean (Standard Deviation); unit: Millimeter
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 38
Number analyzed (Target lesions) | 38
Millimeter | 0.12 (0.36)

61. Secondary Outcome: Proximal Late Loss: Proximal MLD Post-procedure - Proximal MLD at 3 Years
Description: as for outcome 58
Time Frame: 3 years
Population: as for outcome 56
Measure: Mean (Standard Deviation); unit: Millimeter
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 43
Number analyzed (Target lesions) | 44
Millimeter | 0.14 (0.31)

62. Secondary Outcome: Proximal Late Loss: Proximal MLD Post-procedure - Proximal MLD at 5 Years
Description: as for outcome 58
Time Frame: 5 years
Population: Intent-to-treat (ITT) population. In Cohort B, Group 1 and Group 2. The number of participants analyzed include subjects who had available follow-up data at that time frame.
Measure: Mean (Standard Deviation); unit: Millimeter
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 57
Number analyzed (Target lesions) | 58
Millimeter | 0.14 (0.43)

63. Secondary Outcome: Distal Late Loss: Distal MLD Post-procedure - Distal MLD at 180 Days
Description: Distal Late Loss: distal MLD post-procedure - distal MLD at follow-up (distal defined as within 5 mm of healthy tissue distal to scaffold placement).
Time Frame: 180 days
Population: Intent-to-treat (ITT) population. Cohort B, Group 1. The number of participants analyzed include subjects who had available follow-up data at that time frame.
Measure: Mean (Standard Deviation); unit: Millimeter
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 41
Number analyzed (Target lesions) | 41
Millimeter | 0.07 (0.30)

64. Secondary Outcome: Distal Late Loss: Distal MLD Post-procedure - Distal MLD at 1 Year
Description: as for outcome 63
Time Frame: 1 year
Population: Intent-to-treat (ITT) population. Cohort B, Group 2. The number of participants analyzed include subjects who had available follow-up data at that time frame.
Measure: Mean (Standard Deviation); unit: Millimeter
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 54
Number analyzed (Target lesions) | 55
Millimeter | 0.07 (0.27)

65. Secondary Outcome: Distal Late Loss: Distal MLD Post-procedure - Distal MLD at 2 Years
Description: as for outcome 63
Time Frame: 2 years
Population: as for outcome 63
Measure: Mean (Standard Deviation); unit: Millimeter
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 37
Number analyzed (Target lesions) | 37
Millimeter | 0.04 (0.25)

66. Secondary Outcome: Distal Late Loss: Distal MLD Post-procedure - Distal MLD at 3 Years
Description: as for outcome 63
Time Frame: 3 years
Population: as for outcome 64
Measure: Mean (Standard Deviation); unit: Millimeter
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 48
Number analyzed (Target lesions) | 49
Millimeter | 0.08 (0.37)

67. Secondary Outcome: Distal Late Loss: Distal MLD Post-procedure - Distal MLD at 5 Years
Description: as for outcome 63
Time Frame: 5 years
Population: as for outcome 57
Measure: Mean (Standard Deviation); unit: Millimeter
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 60
Number analyzed (Target lesions) | 61
Millimeter | 0.11 (0.35)

68. Secondary Outcome: In-scaffold Angiographic Binary Restenosis (ABR)
Description: Percent of patients with a followup percent diameter stenosis of >=50% per QCA.
Time Frame: 180 days
Population: as for outcome 63
Measure: Number; unit: Percentage of participants
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 42
Number analyzed (Target lesions) | 42
Percentage of participants | 0.0

69. Secondary Outcome: In-scaffold Angiographic Binary Restenosis (ABR)
Description: Percent of patients with a followup percent diameter stenosis of >=50% per QCA.
Time Frame: 1 year
Population: as for outcome 64
Measure: Number; unit: Percentage of participants
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 56
Number analyzed (Target lesions) | 57
Percentage of participants | 3.5

70. Secondary Outcome: In-scaffold Angiographic Binary Restenosis (ABR)
Description: Percent of patients with a followup percent diameter stenosis of >=50% per QCA.
Time Frame: 2 years
Population: as for outcome 63
Measure: Number; unit: Percentage of participants
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 38
Number analyzed (Target lesions) | 38
Percentage of participants | 0.0

71. Secondary Outcome: In-scaffold Angiographic Binary Restenosis (ABR)
Description: Percent of patients with a followup percent diameter stenosis of >=50% per QCA.
Time Frame: 3 years
Population: as for outcome 64
Measure: Number; unit: Percentage of participants
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 50
Number analyzed (Target lesions) | 51
Percentage of participants | 7.8

72. Secondary Outcome: In-scaffold Angiographic Binary Restenosis (ABR)
Description: Percent of patients with a followup percent diameter stenosis of >=50% per QCA.
Time Frame: 5 years
Population: as for outcome 57
Measure: Number; unit: Percentage of participants
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 63
Number analyzed (Target lesions) | 64
Percentage of participants | 7.8

73. Secondary Outcome: Persisting Dissection
Description: Dissection at follow-up that was present post-procedure.
Time Frame: 180 days
Population: ITT population. Cohort B, Group 1. The number of participants analyzed include subjects who had available follow-up data at that time frame.
Measure: Number; unit: Percentage of participants
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 42
Number analyzed (Target lesions) | 42
Percentage of participants | 0.0

74. Secondary Outcome: Persisting Dissection
Description: Dissection at follow-up that was present post-procedure.
Time Frame: 1 year
Population: ITT population. Cohort B, Group 2. The number of participants analyzed include subjects who had available follow-up data at that time frame.
Measure: Number; unit: Percentage of participants
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 56
Number analyzed (Target lesions) | 57
Percentage of participants | 0.0

75. Secondary Outcome: Persisting Dissection
Description: Dissection at follow-up that was present post-procedure.
Time Frame: 2 years
Population: as for outcome 73
Measure: Number; unit: Percentage of participants
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 38
Number analyzed (Target lesions) | 38
Percentage of participants | 0.0

76. Secondary Outcome: Persisting Dissection
Description: Dissection at follow-up that was present post-procedure.
Time Frame: 3 years
Population: as for outcome 74
Measure: Number; unit: Percentage of participants
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 47
Number analyzed (Target lesions) | 48
Percentage of participants | 0.0

77. Secondary Outcome: Persisting Dissection
Description: Dissection at follow-up that was present post-procedure.
Time Frame: 5 years
Population: ITT population. Cohort B, Group 1 and Group 2. The number of participants analyzed include subjects who had available follow-up data at that time frame.
Measure: Number; unit: Percentage of participants
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 47
Number analyzed (Target lesions) | 48
Percentage of participants | 0.0

78. Secondary Outcome: In-scaffold Percent Diameter Stenosis (%DS)
Description: Percent Diameter Stenosis is defined as the value calculated as 100 * (1 - MLD/RVD) using the mean values from two orthogonal views (when possible) by QCA.
Time Frame: 180 days
Population: as for outcome 63
Measure: Mean (Standard Deviation); unit: percentage of diameter stenosis
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 42
Number analyzed (Target lesions) | 42
percentage of diameter stenosis | 19.21 (7.62)

79. Secondary Outcome: In-scaffold Percent Diameter Stenosis (%DS)
Description: as for outcome 78
Time Frame: 1 year
Population: as for outcome 64
Measure: Mean (Standard Deviation); unit: percentage of diameter stenosis
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 55
Number analyzed (Target lesions) | 56
percentage of diameter stenosis | 21.35 (11.18)

80. Secondary Outcome: In-scaffold Percent Diameter Stenosis (%DS)
Description: as for outcome 78
Time Frame: 2 years
Population: as for outcome 63
Measure: Mean (Standard Deviation); unit: percentage of diameter stenosis
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 38
Number analyzed (Target lesions) | 38
percentage of diameter stenosis | 20.94 (7.63)

81. Secondary Outcome: In-scaffold Percent Diameter Stenosis (%DS)
Description: as for outcome 78
Time Frame: 3 years
Population: as for outcome 64
Measure: Mean (Standard Deviation); unit: percentage of diameter stenosis
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 50
Number analyzed (Target lesions) | 51
percentage of diameter stenosis | 23.16 (14.85)

82. Secondary Outcome: In-scaffold Percent Diameter Stenosis (%DS)
Description: as for outcome 78
Time Frame: 5 years
Population: Intent-to-treat (ITT) population. Cohort B, Group 1 and Group2. The number of participants analyzed include subjects who had available follow-up data at that time frame.
Measure: Mean (Standard Deviation); unit: percentage of diameter stenosis
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 63
Number analyzed (Target lesions) | 64
percentage of diameter stenosis | 22.74 (13.94)

83. Secondary Outcome: Aneurysm
Description: An abnormal expansion or protrusion of a coronary blood vessel resulting from a disease or weakening of the vessel's wall (all three layers) that exceeds the RVD of the vessel by 1.5 times.
Time Frame: 180 days
Population: as for outcome 63
Measure: Number; unit: Percentage of participants
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 42
Number analyzed (Target lesions) | 42
Percentage of participants | 2.4

84. Secondary Outcome: Aneurysm
Description: as for outcome 83
Time Frame: 1 year
Population: as for outcome 64
Measure: Number; unit: Percentage of participants
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 56
Number analyzed (Target lesions) | 57
Percentage of participants | 0.0

85. Secondary Outcome: Aneurysm
Description: as for outcome 83
Time Frame: 2 years
Population: as for outcome 63
Measure: Number; unit: Percentage of participants
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 38
Number analyzed (Target lesions) | 38
Percentage of participants | 2.6

86. Secondary Outcome: Aneurysm
Description: as for outcome 83
Time Frame: 3 years
Population: as for outcome 64
Measure: Number; unit: Percentage of participants
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 47
Number analyzed (Target lesions) | 48
Percentage of participants | 2.08

87. Secondary Outcome: Aneurysm
Description: as for outcome 83
Time Frame: 5 years
Population: Intent-to-treat (ITT) population.Cohort B, Group 1 and Group 2. The number of participants analyzed include subjects who had available follow-up data at that time frame.
Measure: Number; unit: Percentage of participants
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 47
Number analyzed (Target lesions) | 48
Percentage of participants | 0.0

88. Secondary Outcome: Thrombus
Time Frame: 180 days
Population: as for outcome 63
Measure: Number; unit: Percentage of participants
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 42
Number analyzed (Target lesions) | 42
Percentage of participants | 0.0

89. Secondary Outcome: Thrombus
Time Frame: 1 year
Population: as for outcome 64
Measure: Number; unit: Percentage of participants
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 56
Number analyzed (Target lesions) | 57
Percentage of participants | 0.0

90. Secondary Outcome: Thrombus
Time Frame: 2 years
Population: Intent-to-treat (ITT) population.Cohort B, Group 1. The number of participants analyzed include subjects who had available follow-up data at that time frame.
Measure: Number; unit: Percentage of participants
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 38
Number analyzed (Target lesions) | 38
Percentage of participants | 2.6

91. Secondary Outcome: Thrombus
Time Frame: 3 years
Population: as for outcome 64
Measure: Number; unit: Percentage of participants
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 47
Number analyzed (Target lesions) | 48
Percentage of participants | 2.08

92. Secondary Outcome: Thrombus
Time Frame: 5 years
Population: as for outcome 57
Measure: Number; unit: Percentage of participants
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 47
Number analyzed (Target lesions) | 48
Percentage of participants | 0.0

93. Secondary Outcome: Vasomotion Analysis: In-scaffold Mean Luminal Diameter
Description: Vasomotion function was assessed in reaction to nitrate administration.
Time Frame: 5 years
Population: Intent-to-treat (ITT) population. The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: Millimeter
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 52
Number analyzed (Target lesions) | 57
Millimeter
  Pre-Nitro | 2.49 (0.37)
  Post-Nitro | 2.56 (0.35)

94. Secondary Outcome: Volume Obstruction (VO)
Description: Defined as scaffold intimal hyperplasia and calculated as 100*(Scaffold Volume - Lumen Volume)/Scaffold Volume by IVUS.
Time Frame: 180 days
Population: Cohort B, Group 1. ITT population; Intravascular ultrasound (IVUS) analysis. The number of participants analyzed include subjects who had available follow-up data at that time frame.
Measure: Mean (Standard Deviation); unit: percent of scaffold volume
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 40
Number analyzed (Target lesions) | 40
percent of scaffold volume | 1.22 (1.99)

95. Secondary Outcome: Volume Obstruction (VO)
Description: Defined as scaffold intimal hyperplasia and calculated as 100*(Scaffold Volume - Lumen Volume)/Scaffold Volume by IVUS.
Time Frame: 1 year
Population: Cohort B, Group 2. ITT population; IVUS analysis. The number of participants analyzed include subjects who had available follow-up data at that time frame.
Measure: Mean (Standard Deviation); unit: percent of scaffold volume
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 55
Number analyzed (Target lesions) | 56
percent of scaffold volume | 1.47 (3.08)

96. Secondary Outcome: Volume Obstruction (VO)
Description: Defined as scaffold intimal hyperplasia and calculated as 100*(Scaffold Volume - Lumen Volume)/Scaffold Volume by IVUS.
Time Frame: 2 year
Population: Cohort B, Group 1. ITT population; IVUS analysis. The number of participants analyzed include subjects who had available follow-up data at that time frame.
Measure: Mean (Standard Deviation); unit: percent of scaffold volume
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 38
Number analyzed (Target lesions) | 38
percent of scaffold volume | 3.33 (3.99)

97. Secondary Outcome: Volume Obstruction (VO)
Description: Defined as scaffold intimal hyperplasia and calculated as 100*(Scaffold Volume - Lumen Volume)/Scaffold Volume by IVUS.
Time Frame: 3 year
Population: as for outcome 95
Measure: Mean (Standard Deviation); unit: percent of scaffold volume
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 45
Number analyzed (Target lesions) | 46
percent of scaffold volume | 4.19 (6.43)

98. Secondary Outcome: Persisting Incomplete Apposition
Description: Persisting incomplete apposition is defined as incomplete apposition at follow-up that was present post-procedure.
  Incomplete Apposition: Failure of the scaffold to completely appose to the vessel wall after placement is defined as one or more scaffold strut separated from the vessel wall with evidence of blood speckles behind the strut in the ultrasound image.
Time Frame: 180 days
Population: Cohort B, Group 1. Intent-to-treat (ITT) population. The number of participants analyzed include subjects who had available follow-up data at that time frame.
Measure: Number; unit: Percentage of participants
Arm/Group | Absorb BVS
Number analyzed (Participants) | 43
Percentage of participants | 2.3

99. Secondary Outcome: Persisting Incomplete Apposition
Description: as for outcome 98
Time Frame: 1 year
Population: Cohort B, Group 2. Intent-to-treat (ITT) population. The number of participants analyzed include subjects who had available follow-up data at that time frame.
Measure: Number; unit: Percentage of participants
Arm/Group | Absorb BVS
Number analyzed (Participants) | 57
Percentage of participants | 3.5

100. Secondary Outcome: Persisting Incomplete Apposition
Description: as for outcome 98
Time Frame: 2 year
Population: as for outcome 98
Measure: Number; unit: Percentage of participants
Arm/Group | Absorb BVS
Number analyzed (Participants) | 43
Percentage of participants | 0.0

101. Secondary Outcome: Persisting Incomplete Apposition
Description: as for outcome 98
Time Frame: 3 year
Population: as for outcome 99
Measure: Number; unit: Percentage of participants
Arm/Group | Absorb BVS
Number analyzed (Participants) | 49
Percentage of participants | 0.0

102. Secondary Outcome: Late Incomplete Apposition
Description: Late-Acquired Incomplete Apposition is defined as incomplete apposition of the scaffold at follow-up, which was not present post-procedure.
  Incomplete Apposition: Failure of the scaffold to completely appose to the vessel wall after placement is defined as one or more scaffold strut separated from the vessel wall with evidence of blood speckles behind the strut in the ultrasound image.
Time Frame: 180 days
Population: as for outcome 98
Measure: Number; unit: Percentage of participants
Arm/Group | Absorb BVS
Number analyzed (Participants) | 40
Percentage of participants | 7.5

103. Secondary Outcome: Late Incomplete Apposition
Description: as for outcome 102
Time Frame: 1 year
Population: as for outcome 99
Measure: Number; unit: Percentage of participants
Arm/Group | Absorb BVS
Number analyzed (Participants) | 56
Percentage of participants | 3.6

104. Secondary Outcome: Late Incomplete Apposition
Description: as for outcome 102
Time Frame: 2 year
Population: as for outcome 98
Measure: Number; unit: Percentage of participants
Arm/Group | Absorb BVS
Number analyzed (Participants) | 38
Percentage of participants | 2.6

105. Secondary Outcome: Late Incomplete Apposition
Description: as for outcome 102
Time Frame: 3 year
Population: as for outcome 99
Measure: Number; unit: Percentage of participants
Arm/Group | Absorb BVS
Number analyzed (Participants) | 43
Percentage of participants | 7.0

106. Other Pre Specified Outcome: Mean Reference Area
Time Frame: 1 year
Population: Optical coherence tomography (OCT) analysis,Cohort B Group 2, Intent-to-Treat Population. The number of participants analyzed include subjects who had available follow-up data at that time frame.
Measure: Mean (Standard Deviation); unit: mm^2
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 30
Number analyzed (Target lesions) | 31
mm^2 | 6.34 (2.30)

107. Other Pre Specified Outcome: Mean Reference Area
Time Frame: 2 years
Population: OCT analysis,Cohort B Group1 , Intent-to-Treat Population. The number of participants analyzed include subjects who had available follow-up data at that time frame.
Measure: Mean (Standard Deviation); unit: mm^2
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 26
Number analyzed (Target lesions) | 27
mm^2 | 6.29 (2.13)

108. Other Pre Specified Outcome: Mean Reference Area
Time Frame: 3 years
Population: OCT analysis,Cohort B Group 2, Intent-to-Treat Population. The number of participants analyzed include subjects who had available follow-up data at that time frame.
Measure: Mean (Standard Deviation); unit: mm^2
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 39
Number analyzed (Target lesions) | 40
mm^2 | 6.24 (1.78)

109. Other Pre Specified Outcome: Mean Reference Area
Time Frame: 5 years
Population: OCT analysis,Cohort B (Group 1 and Group 2), Intent-to-Treat Population. The number of participants analyzed include subjects who had available follow-up data at that time frame.
Measure: Mean (Standard Deviation); unit: mm^2
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 49
Number analyzed (Target lesions) | 50
mm^2 | 6.13 (1.96)

110. Other Pre Specified Outcome: Mean Luminal Area
Time Frame: 1 year
Population: Cohort B Group 2, Intent-to-Treat Population. OCT analysis. The number of participants analyzed include subjects who had available follow-up data at that time frame.
Measure: Mean (Standard Deviation); unit: mm^2
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 31
Number analyzed (Target lesions) | 31
mm^2 | 5.92 (1.71)

111. Other Pre Specified Outcome: Mean Luminal Area
Time Frame: 2 years
Population: Cohort B Group 1, Intent-to-Treat Population. OCT analysis. The number of participants analyzed include subjects who had available follow-up data at that time frame.
Measure: Mean (Standard Deviation); unit: mm^2
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 27
Number analyzed (Target lesions) | 28
mm^2 | 6.00 (1.76)

112. Other Pre Specified Outcome: Mean Luminal Area
Time Frame: 3 years
Population: as for outcome 110
Measure: Mean (Standard Deviation); unit: mm^2
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 45
Number analyzed (Target lesions) | 45
mm^2 | 6.06 (1.70)

113. Other Pre Specified Outcome: Mean Luminal Area
Time Frame: 5 years
Population: Cohort B (Group 1 and Group 2), Intent-to-Treat (ITT) Population.OCT analysis. The number of participants analyzed include subjects who had available follow-up data at that time frame.
Measure: Mean (Standard Deviation); unit: mm^2
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 53
Number analyzed (Target lesions) | 54
mm^2 | 6.22 (1.84)

114. Other Pre Specified Outcome: Minimum Luminal Area
Time Frame: 1 year
Population: as for outcome 110
Measure: Mean (Standard Deviation); unit: mm^2
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 31
Number analyzed (Target lesions) | 31
mm^2 | 4.29 (1.39)

115. Other Pre Specified Outcome: Minimum Luminal Area
Time Frame: 2 years
Population: as for outcome 111
Measure: Mean (Standard Deviation); unit: mm^2
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 27
Number analyzed (Target lesions) | 28
mm^2 | 4.29 (1.48)

116. Other Pre Specified Outcome: Minimum Luminal Area
Time Frame: 3 years
Population: as for outcome 110
Measure: Mean (Standard Deviation); unit: mm^2
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 45
Number analyzed (Target lesions) | 45
mm^2 | 4.45 (1.55)

117. Other Pre Specified Outcome: Minimum Luminal Area
Time Frame: 5 years
Population: Cohort B (Group 1 and Group 2), Intent-to-Treat Population. OCT analysis. The number of participants analyzed include subjects who had available follow-up data at that time frame.
Measure: Mean (Standard Deviation); unit: mm^2
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 53
Number analyzed (Target lesions) | 54
mm^2 | 4.15 (1.69)

118. Other Pre Specified Outcome: Mean Stent Area
Time Frame: 1 year
Population: as for outcome 110
Measure: Mean (Standard Deviation); unit: mm^2
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 31
Number analyzed (Target lesions) | 31
mm^2 | 7.42 (1.22)

119. Other Pre Specified Outcome: Mean Scaffold Area
Time Frame: 2 years
Population: as for outcome 111
Measure: Mean (Standard Deviation); unit: mm^2
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 27
Number analyzed (Target lesions) | 28
mm^2 | 8.14 (1.88)

120. Other Pre Specified Outcome: Mean Scaffold Area
Time Frame: 3 years
Population: as for outcome 110
Measure: Mean (Standard Deviation); unit: mm^2
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 45
Number analyzed (Target lesions) | 45
mm^2 | 8.50 (1.93)

121. Other Pre Specified Outcome: Minimum Stent Area
Time Frame: 1 year
Population: as for outcome 110
Measure: Mean (Standard Deviation); unit: mm^2
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 31
Number analyzed (Target lesions) | 31
mm^2 | 5.96 (1.14)

122. Other Pre Specified Outcome: Minimum Scaffold Area
Time Frame: 2 year
Population: as for outcome 111
Measure: Mean (Standard Deviation); unit: mm^2
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 27
Number analyzed (Target lesions) | 28
mm^2 | 6.33 (1.45)

123. Other Pre Specified Outcome: Minimum Scaffold Area
Time Frame: 3 years
Population: as for outcome 110
Measure: Mean (Standard Deviation); unit: mm^2
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 45
Number analyzed (Target lesions) | 45
mm^2 | 6.66 (1.67)

124. Other Pre Specified Outcome: Luminal Volume
Time Frame: 1 year
Population: as for outcome 110
Measure: Mean (Standard Deviation); unit: mm^3
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 31
Number analyzed (Target lesions) | 31
mm^3 | 106.33 (31.42)

125. Other Pre Specified Outcome: Luminal Volume
Time Frame: 2 years
Population: as for outcome 111
Measure: Mean (Standard Deviation); unit: mm^3
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 27
Number analyzed (Target lesions) | 28
mm^3 | 107.66 (34.79)

126. Other Pre Specified Outcome: Luminal Volume
Time Frame: 3 years
Population: as for outcome 110
Measure: Mean (Standard Deviation); unit: mm^3
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 45
Number analyzed (Target lesions) | 45
mm^3 | 103.31 (30.86)

127. Other Pre Specified Outcome: Luminal Volume
Time Frame: 5 years
Population: Cohort B Group 1 and Group 2, Intent-to-Treat Population. OCT analysis. The number of participants analyzed include subjects who had available follow-up data at that time frame.
Measure: Mean (Standard Deviation); unit: mm^3
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 53
Number analyzed (Target lesions) | 54
mm^3 | 106.36 (32.72)

128. Other Pre Specified Outcome: Stent Volume
Time Frame: 1 year
Population: as for outcome 110
Measure: Mean (Standard Deviation); unit: mm^3
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 31
Number analyzed (Target lesions) | 31
mm^3 | 132.90 (21.64)

129. Other Pre Specified Outcome: Scaffold Volume
Time Frame: 2 years
Population: as for outcome 111
Measure: Mean (Standard Deviation); unit: mm^3
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 27
Number analyzed (Target lesions) | 28
mm^3 | 145.78 (38.28)

130. Other Pre Specified Outcome: Scaffold Volume
Time Frame: 3 years
Population: as for outcome 110
Measure: Mean (Standard Deviation); unit: mm^3
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 45
Number analyzed (Target lesions) | 45
mm^3 | 145.07 (36.69)

131. Other Pre Specified Outcome: Mean Luminal Diameter
Time Frame: 1 year
Population: as for outcome 110
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 31
Number analyzed (Target lesions) | 31
mm | 2.71 (0.39)

132. Other Pre Specified Outcome: Mean Luminal Diameter
Time Frame: 2 years
Population: as for outcome 111
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 27
Number analyzed (Target lesions) | 28
mm | 2.72 (0.42)

133. Other Pre Specified Outcome: Mean Luminal Diameter
Time Frame: 3 years
Population: as for outcome 110
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 45
Number analyzed (Target lesions) | 45
mm | 2.74 (0.39)

134. Other Pre Specified Outcome: Mean Luminal Diameter
Description: It is measured during QCA by the Angiographic Core Lab.
Time Frame: 5 years
Population: as for outcome 117
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 53
Number analyzed (Target lesions) | 54
mm | 2.77 (0.42)

135. Other Pre Specified Outcome: Minimum Luminal Diameter (MLD)
Description: The average of two orthogonal views (when possible) of the narrowest point within the area of assessment - in lesion, in scaffold or in segment. MLD is visually estimated during angiography by the Investigator; it is measured during QCA by the Angiographic Core Lab.
Time Frame: 1 year
Population: as for outcome 110
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 31
Number analyzed (Target lesions) | 31
mm | 2.30 (0.42)

136. Other Pre Specified Outcome: Minimum Luminal Diameter
Description: as for outcome 135
Time Frame: 2 years
Population: Cohort B Group 1 , Intent-to-Treat Population. OCT analysis. The number of participants analyzed include subjects who had available follow-up data at that time frame.
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 27
Number analyzed (Target lesions) | 28
mm | 2.30 (0.40)

137. Other Pre Specified Outcome: Minimum Luminal Diameter
Description: as for outcome 135
Time Frame: 3 years
Population: as for outcome 110
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 45
Number analyzed (Target lesions) | 45
mm | 2.34 (0.46)

138. Other Pre Specified Outcome: Minimum Luminal Diameter
Description: as for outcome 135
Time Frame: 5 years
Population: Cohort B (Group1 and Group 2), Intent-to-Treat Population. OCT analysis. The number of participants analyzed include subjects who had available follow-up data at that time frame.
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 53
Number analyzed (Target lesions) | 54
mm | 2.25 (0.49)

139. Other Pre Specified Outcome: Mean Stent Diameter
Time Frame: 1 year
Population: as for outcome 110
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 31
Number analyzed (Target lesions) | 31
mm | 3.06 (0.24)

140. Other Pre Specified Outcome: Mean Scaffold Diameter
Time Frame: 2 years
Population: as for outcome 111
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 27
Number analyzed (Target lesions) | 28
mm | 3.19 (0.38)

141. Other Pre Specified Outcome: Mean Scaffold Diameter
Time Frame: 3 years
Population: as for outcome 110
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 45
Number analyzed (Target lesions) | 45
mm | 3.26 (0.36)

142. Other Pre Specified Outcome: Minimum Stent Diameter
Time Frame: 1 year
Population: as for outcome 110
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 31
Number analyzed (Target lesions) | 31
mm | 2.74 (0.26)

143. Other Pre Specified Outcome: Minimum Scaffold Diameter
Time Frame: 2 years
Population: as for outcome 111
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 27
Number analyzed (Target lesions) | 28
mm | 2.82 (0.33)

144. Other Pre Specified Outcome: Minimum Scaffold Diameter
Time Frame: 3 years
Population: as for outcome 110
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 45
Number analyzed (Target lesions) | 45
mm | 2.89 (0.37)

145. Other Pre Specified Outcome: Strut Volume
Time Frame: 1 year
Population: as for outcome 110
Measure: Mean (Standard Deviation); unit: mm^3
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 31
Number analyzed (Target lesions) | 31
mm^3 | 3.02 (0.66)

146. Other Pre Specified Outcome: Strut Volume
Time Frame: 2 years
Population: as for outcome 111
Measure: Mean (Standard Deviation); unit: mm^3
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 27
Number analyzed (Target lesions) | 28
mm^3 | 2.61 (0.45)

147. Other Pre Specified Outcome: Strut Volume
Time Frame: 3 years
Population: as for outcome 110
Measure: Mean (Standard Deviation); unit: mm^3
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 45
Number analyzed (Target lesions) | 45
mm^3 | 3.28 (0.83)

148. Other Pre Specified Outcome: Number of Struts Per BVS
Time Frame: 1 year
Population: as for outcome 110
Measure: Mean (Standard Deviation); unit: Number of Struts
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 30
Number analyzed (Target lesions) | 31
Number of Struts | 162.1 (31.9)

149. Other Pre Specified Outcome: Number of Struts Per BVS
Time Frame: 2 years
Population: as for outcome 111
Measure: Mean (Standard Deviation); unit: Number of Struts
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 27
Number analyzed (Target lesions) | 28
Number of Struts | 160.9 (27.9)

150. Other Pre Specified Outcome: Number of Struts Per BVS
Time Frame: 3 years
Population: as for outcome 110
Measure: Mean (Standard Deviation); unit: Number of Struts
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 45
Number analyzed (Target lesions) | 45
Number of Struts | 145.2 (32.3)

151. Other Pre Specified Outcome: Number of Struts Per BVS
Time Frame: 5 years
Population: as for outcome 117
Measure: Mean (Standard Deviation); unit: Number of Struts
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 53
Number analyzed (Target lesions) | 54
Number of Struts | 7.1 (29.1)

152. Other Pre Specified Outcome: % of Covered Struts (150 µm)
Time Frame: 1 year
Population: as for outcome 110
Measure: Mean (Standard Deviation); unit: Percent of Covered Struts
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 31
Number analyzed (Target lesions) | 31
Percent of Covered Struts | 96.86 (2.95)

153. Other Pre Specified Outcome: % of Acutely Covered Struts
Time Frame: 2 years
Population: as for outcome 111
Measure: Mean (Standard Deviation); unit: Percent of Covered Struts
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 27
Number analyzed (Target lesions) | 28
Percent of Covered Struts | 98.07 (3.27)

154. Other Pre Specified Outcome: % of Acutely Covered Struts
Time Frame: 3 years
Population: as for outcome 110
Measure: Mean (Standard Deviation); unit: Percent of Covered Struts
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 45
Number analyzed (Target lesions) | 45
Percent of Covered Struts | 97.90 (2.00)

155. Other Pre Specified Outcome: % of Uncovered Struts (150 µm)
Time Frame: 1 year
Population: as for outcome 110
Measure: Mean (Standard Deviation); unit: Percent of Uncovered Struts
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 31
Number analyzed (Target lesions) | 31
Percent of Uncovered Struts | 3.14 (2.95)

156. Other Pre Specified Outcome: % of Uncovered Struts (150 µm)
Time Frame: 2 years
Population: as for outcome 111
Measure: Mean (Standard Deviation); unit: Percent of Uncovered Struts
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 27
Number analyzed (Target lesions) | 28
Percent of Uncovered Struts | 1.93 (3.27)

157. Other Pre Specified Outcome: % of Uncovered Struts (150 µm)
Time Frame: 3 years
Population: as for outcome 110
Measure: Mean (Standard Deviation); unit: Percent of Uncovered Struts
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 45
Number analyzed (Target lesions) | 45
Percent of Uncovered Struts | 2.10 (2.00)

158. Other Pre Specified Outcome: Number of Struts in Side Branch
Time Frame: 1 year
Population: as for outcome 110
Measure: Mean (Standard Deviation); unit: Number of struts
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 31
Number analyzed (Target lesions) | 31
Number of struts | 0.1 (0.4)

159. Other Pre Specified Outcome: Number of Struts in Side Branch
Time Frame: 2 years
Population: as for outcome 111
Measure: Mean (Standard Deviation); unit: Number of struts
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 27
Number analyzed (Target lesions) | 28
Number of struts | 0.2 (0.6)

160. Other Pre Specified Outcome: Number of Struts in Side Branch
Time Frame: 3 years
Population: as for outcome 110
Measure: Mean (Standard Deviation); unit: Number of struts
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 45
Number analyzed (Target lesions) | 45
Number of struts | 0.2 (0.4)

161. Other Pre Specified Outcome: Number of Struts in Side Branch
Time Frame: 5 years
Population: as for outcome 117
Measure: Mean (Standard Deviation); unit: Number of struts
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 53
Number analyzed (Target lesions) | 54
Number of struts | 0.0 (0.3)

162. Other Pre Specified Outcome: Tissue Coverage Area Classical
Time Frame: 1 year
Population: as for outcome 110
Measure: Mean (Standard Deviation); unit: mm^2
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 31
Number analyzed (Target lesions) | 31
mm^2 | 1.54 (0.76)

163. Other Pre Specified Outcome: Tissue Coverage Area BVS (Neointimal Area)
Time Frame: 1 year
Population: as for outcome 110
Measure: Mean (Standard Deviation); unit: mm^2
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 27
Number analyzed (Target lesions) | 31
mm^2 | 1.38 (0.75)

164. Other Pre Specified Outcome: Tissue Coverage Volume Classical
Time Frame: 1 year
Population: as for outcome 110
Measure: Mean (Standard Deviation); unit: mm^3
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 31
Number analyzed (Target lesions) | 31
mm^3 | 27.27 (13.16)

165. Other Pre Specified Outcome: Tissue Coverage Volume BVS
Time Frame: 1 year
Population: as for outcome 110
Measure: Mean (Standard Deviation); unit: mm^3
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 31
Number analyzed (Target lesions) | 31
mm^3 | 24.40 (12.97)

166. Other Pre Specified Outcome: Tissue Coverage Obstruction Volume Classical
Time Frame: 1 year
Population: as for outcome 110
Measure: Mean (Standard Deviation); unit: Percent of Tissue Coverage Obstruction
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 31
Number analyzed (Target lesions) | 31
Percent of Tissue Coverage Obstruction | 21.61 (11.77)

167. Other Pre Specified Outcome: Tissue Coverage Obstruction Volume BVS
Time Frame: 1 year
Population: as for outcome 110
Measure: Mean (Standard Deviation); unit: Percent of Tissue Coverage Obstruction
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 31
Number analyzed (Target lesions) | 31
Percent of Tissue Coverage Obstruction | 19.40 (11.52)

168. Other Pre Specified Outcome: Tissue Coverage Area Classical
Time Frame: 2 years
Population: as for outcome 111
Measure: Mean (Standard Deviation); unit: mm^2
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 27
Number analyzed (Target lesions) | 28
mm^2 | 2.13 (0.58)

169. Other Pre Specified Outcome: Tissue Coverage Area BVS (Neointimal Area)
Time Frame: 2 years
Population: as for outcome 111
Measure: Mean (Standard Deviation); unit: mm^2
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 27
Number analyzed (Target lesions) | 28
mm^2 | 1.99 (0.58)

170. Other Pre Specified Outcome: Tissue Coverage Volume Classical
Time Frame: 2 years
Population: as for outcome 111
Measure: Mean (Standard Deviation); unit: mm^3
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 27
Number analyzed (Target lesions) | 28
mm^3 | 38.12 (10.99)

171. Other Pre Specified Outcome: Tissue Coverage Volume BVS
Time Frame: 2 years
Population: as for outcome 111
Measure: Mean (Standard Deviation); unit: mm^3
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 27
Number analyzed (Target lesions) | 28
mm^3 | 35.51 (10.87)

172. Other Pre Specified Outcome: Tissue Coverage Obstruction Volume Classical
Time Frame: 2 years
Population: as for outcome 111
Measure: Mean (Standard Deviation); unit: Percent of Tissue Coverage Obstruction
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 27
Number analyzed (Target lesions) | 28
Percent of Tissue Coverage Obstruction | 27.10 (8.16)

173. Other Pre Specified Outcome: Tissue Coverage Obstruction Volume BVS
Time Frame: 2 years
Population: as for outcome 111
Measure: Mean (Standard Deviation); unit: Percent of Tissue Coverage Obstruction
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 27
Number analyzed (Target lesions) | 28
Percent of Tissue Coverage Obstruction | 25.22 (7.91)

174. Other Pre Specified Outcome: Tissue Coverage Area Classical
Time Frame: 3 years
Population: as for outcome 110
Measure: Mean (Standard Deviation); unit: mm^2
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 45
Number analyzed (Target lesions) | 45
mm^2 | 2.44 (0.61)

175. Other Pre Specified Outcome: Tissue Coverage Area BVS (Neointimal Area)
Time Frame: 3 years
Population: as for outcome 110
Measure: Mean (Standard Deviation); unit: mm^2
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 45
Number analyzed (Target lesions) | 45
mm^2 | 2.25 (0.60)

176. Other Pre Specified Outcome: Tissue Coverage Volume Classical
Time Frame: 3 years
Population: as for outcome 110
Measure: Mean (Standard Deviation); unit: mm^3
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 45
Number analyzed (Target lesions) | 45
mm^3 | 41.76 (11.46)

177. Other Pre Specified Outcome: Tissue Coverage Volume BVS
Time Frame: 3 years
Population: as for outcome 110
Measure: Mean (Standard Deviation); unit: mm^3
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 45
Number analyzed (Target lesions) | 45
mm^3 | 38.47 (11.20)

178. Other Pre Specified Outcome: Tissue Coverage Obstruction Volume Classical
Time Frame: 3 years
Population: as for outcome 110
Measure: Mean (Standard Deviation); unit: Percent of Tissue Coverage Obstruction
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 45
Number analyzed (Target lesions) | 45
Percent of Tissue Coverage Obstruction | 29.36 (7.28)

179. Other Pre Specified Outcome: Tissue Coverage Obstruction Volume BVS
Time Frame: 3 years
Population: as for outcome 110
Measure: Mean (Standard Deviation); unit: Percent of Tissue Coverage Obstruction
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 45
Number analyzed (Target lesions) | 45
Percent of Tissue Coverage Obstruction | 27.01 (7.10)

180. Other Pre Specified Outcome: Mean Flow Area
Time Frame: 1 year
Population: as for outcome 110
Measure: Mean (Standard Deviation); unit: mm^2
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 31
Number analyzed (Target lesions) | 31
mm^2 | 5.90 (1.66)

181. Other Pre Specified Outcome: Minimum Flow Area
Time Frame: 1 year
Population: as for outcome 110
Measure: Mean (Standard Deviation); unit: mm^2
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 31
Number analyzed (Target lesions) | 31
mm^2 | 4.28 (1.39)

182. Other Pre Specified Outcome: Mean Strut Core Area
Time Frame: 1 year
Population: as for outcome 110
Measure: Mean (Standard Deviation); unit: mm^2
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 31
Number analyzed (Target lesions) | 31
mm^2 | 0.17 (0.05)

183. Other Pre Specified Outcome: Percent (%) Lumen Area Stenosis
Time Frame: 1 year
Population: as for outcome 110
Measure: Mean (Standard Deviation); unit: Percentage of Lumen Area Stenosis
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 31
Number analyzed (Target lesions) | 31
Percentage of Lumen Area Stenosis | 28.70 (12.05)

184. Other Pre Specified Outcome: Mean Flow Area
Time Frame: 2 years
Population: as for outcome 111
Measure: Mean (Standard Deviation); unit: mm^2
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 27
Number analyzed (Target lesions) | 28
mm^2 | 6.00 (1.76)

185. Other Pre Specified Outcome: Minimum Flow Area
Time Frame: 2 years
Population: as for outcome 111
Measure: Mean (Standard Deviation); unit: mm^2
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 27
Number analyzed (Target lesions) | 28
mm^2 | 4.29 (1.47)

186. Other Pre Specified Outcome: Mean Strut Core Area
Time Frame: 2 years
Population: as for outcome 111
Measure: Mean (Standard Deviation); unit: mm^2
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 27
Number analyzed (Target lesions) | 28
mm^2 | 0.15 (0.02)

187. Other Pre Specified Outcome: Percent (%) Lumen Area Stenosis
Time Frame: 2 years
Population: as for outcome 111
Measure: Mean (Standard Deviation); unit: Percentage of Lumen Area Stenosis
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 27
Number analyzed (Target lesions) | 28
Percentage of Lumen Area Stenosis | 28.75 (10.58)

188. Other Pre Specified Outcome: Mean Flow Area
Time Frame: 3 years
Population: as for outcome 110
Measure: Mean (Standard Deviation); unit: mm^2
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 45
Number analyzed (Target lesions) | 45
mm^2 | 6.06 (1.70)

189. Other Pre Specified Outcome: Minimum Flow Area
Time Frame: 3 years
Population: as for outcome 110
Measure: Mean (Standard Deviation); unit: mm^2
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 45
Number analyzed (Target lesions) | 45
mm^2 | 4.45 (1.55)

190. Other Pre Specified Outcome: Mean Strut Core Area
Time Frame: 3 years
Population: as for outcome 110
Measure: Mean (Standard Deviation); unit: mm^2
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 45
Number analyzed (Target lesions) | 45
mm^2 | 0.19 (0.04)

191. Other Pre Specified Outcome: Percent (%) Lumen Area Stenosis
Time Frame: 3 years
Population: as for outcome 110
Measure: Mean (Standard Deviation); unit: Percentage of Lumen Area Stenosis
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 45
Number analyzed (Target lesions) | 45
Percentage of Lumen Area Stenosis | 28.01 (13.68)

192. Other Pre Specified Outcome: Mean Flow Area
Time Frame: 5 years
Population: as for outcome 117
Measure: Mean (Standard Deviation); unit: mm^2
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 53
Number analyzed (Target lesions) | 54
mm^2 | 6.21 (1.83)

193. Other Pre Specified Outcome: Minimum Flow Area
Time Frame: 5 years
Population: as for outcome 117
Measure: Mean (Standard Deviation); unit: mm^2
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 53
Number analyzed (Target lesions) | 54
mm^2 | 4.15 (1.69)

194. Other Pre Specified Outcome: Percent (%) Lumen Area Stenosis
Time Frame: 5 years
Population: as for outcome 117
Measure: Mean (Standard Deviation); unit: Percentage of Lumen Area Stenosis
Units Other Than Participants: Target lesions
Arm/Group | Absorb BVS
Number analyzed (Participants) | 53
Number analyzed (Target lesions) | 54
Percentage of Lumen Area Stenosis | 34.32 (16.21)

ADVERSE EVENTS:
Time Frame: 5 years
Description: The data for adverse event reporting & clinical outcomes was collected from the full Cohort B (101 patients) up to 5 years (i.e. At Discharge,30 days,270 days,12 months,18 months,2,3,4 & 5 years).The subjects were only divided to Group 1 (n = 45; followed for 6 months, 2 & 5 years) and Group 2 (n = 56; followed for 1, 2 & 5 years) for analyzing imaging outcomes (Angiography, IVUS, Intravascular Ultrasound-virtual histology (IVUS-VH) and OCT imaging procedures) at different follow-up periods.
Arm/Group | ABSORB Stent
All-Cause Mortality (participants affected / at risk) | 0/101
Serious Adverse Events (participants affected / at risk) | 56/101
Other Adverse Events (participants affected / at risk) | 58/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ABSORB Stent (N=101)
Angina pectoris (Cardiac disorders) | 24 (40)
Atrial fibrillation (Cardiac disorders) | 4 (4)
Atrial flutter (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 1 (1)
Coronary artery thrombosis (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 3 (3)
Myocardial ischaemia (Cardiac disorders) | 6 (6)
Palpitations (Cardiac disorders) | 2 (2)
Tachycardia (Cardiac disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2)
Crohn's disease (Gastrointestinal disorders) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Tooth disorder (Gastrointestinal disorders) | 1 (1)
Adverse drug reaction (General disorders) | 1 (1)
Chest discomfort (General disorders) | 1 (1)
Chest pain (General disorders) | 2 (2)
Influenza like illness (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (11)
Thrombosis in device (General disorders) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1)
Bronchopneumonia (Infections and infestations) | 1 (1)
Gangrene (Infections and infestations) | 1 (1)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1)
In-stent coronary artery restenosis (Injury, poisoning and procedural complications) | 1 (1)
Meniscus lesion (Injury, poisoning and procedural complications) | 1 (1)
Cardiac stress test abnormal (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1)
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Carotid artery disease (Nervous system disorders) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 2 (2)
Syncope (Nervous system disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 (3)
Haematoma (Vascular disorders) | 1 (1)
Intermittent claudication (Vascular disorders) | 1 (2)
Varicose vein (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ABSORB Stent (N=101)
Angina pectoris (Cardiac disorders) | 44 (84)
Atrial fibrillation (Cardiac disorders) | 6 (10)
Coronary artery dissection (Cardiac disorders) | 10 (10)
Myocardial ischaemia (Cardiac disorders) | 6 (6)
Non-cardiac chest pain (General disorders) | 18 (30)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 (11)
Haematoma (Vascular disorders) | 8 (8)
Hypertension (Vascular disorders) | 9 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less